CLINICAL TRIAL: NCT02886702
Title: A Multi-Center, Double-Blind, Randomized, Vehicle-Controlled, Parallel-Group Study Comparing Tazarotene Cream 0.05% to TAZORAC® (Tazarotene) Cream 0.05% and Both Active Treatments to a Vehicle Control in the Treatment of Stable Plaque Psoriasis
Brief Title: A Study Comparing Tazarotene Cream 0.05% to TAZORAC® (Tazarotene) Cream 0.05% and Both to a Placebo Control in the Treatment of Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fougera Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0453-01-01; 0453 (Other: Fougera Pharmaceuticals Inc.)
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Results first posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-07

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — tazarotene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test (Experimental): Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.)
  Interventions: Drug: Tazarotene Cream 0.05%
- Reference (Active Comparator): TAZORAC® (tazarotene) Cream 0.05% (Allergan, Inc.)
  Interventions: Drug: TAZORAC® (tazarotene) Cream 0.05%
- Placebo (Placebo Comparator): Placebo (Vehicle of test product) (Fougera Pharmaceuticals Inc.)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tazarotene Cream 0.05% — Tazarotene Cream 0.05% to cover only the lesions with a thin film.
  Other Names: Tazarotene
  Arms: Test
Drug: TAZORAC® (tazarotene) Cream 0.05% — TAZORAC® (tazarotene) Cream 0.05% to cover only the lesions with a thin film.
  Other Names: Tazarotene
  Arms: Reference
Drug: Placebo — Placebo (vehicle of the test product) to cover only the lesions with a thin film.
  Other Names: Vehicle
  Arms: Placebo

SUMMARY:
A Multi-Center, Double-Blind, Randomized, Vehicle-Controlled, Parallel-Group Study Comparing Tazarotene Cream 0.05% to TAZORAC® (tazarotene) Cream 0.05% and Both Active Treatments to a Vehicle Control in the Treatment of Stable Plaque Psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Have a definite clinical diagnosis of stable (at least 6 months) plaque psoriasis, involving at least 2% and no more than 20% of the body surface area (BSA) (not including the scalp and intertriginous areas)
* Have a minimum plaque elevation at the target lesion site of at least moderate severity (grade ≥ 3 on the Psoriasis Area Severity Index [PASI]). The most severe lesion at baseline should be identified as the target lesion
* Have an Investigator's Global Assessment (IGA) of disease severity of at least moderate (score ≥ 3) as an overall assessment of all lesions to be treated.

Exclusion Criteria:

* A female subject who is pregnant, nursing, planning a pregnancy, or does not agree to use an acceptable form of birth control within the study participation period
* Have a current diagnosis of unstable forms of psoriasis in the treatment area, including pustular, guttate, exfoliative or erythrodermic psoriasis
* Have a history of psoriasis unresponsive to topical treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 855 (Actual)
Dates: Start 2016-09-19 (Actual); Primary Completion 2017-08-02 (Actual); Study Completion 2017-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela C. Kaplan, Study Director — Fougera Pharmaceuticals Inc.
Locations (28):
- United States (28):
  - Fougera Investigational Site, Phoenix, Arizona
  - Fougera Investigational Site, Hot Springs, Arkansas
  - Fougera Investigational Site, Anaheim, California
  - Fougera Investigational Site, North Hollywood, California
  - Fougera Investigational Site, San Diego, California
  - Fougera Investigational Site, San Ramon, California
  - Fougera Investigational Site, Brandon, Florida
  - Fougera Investigational Site, Coral Gables, Florida
  - Fougera Investigational Site, Hialeah, Florida
  - Fougera Investigational Site, Miami, Florida
  - Fougera Investigational Site, Miami Gardens, Florida
  - Fougera Investigational Site, Miramar, Florida
  - Fougera Investigational Site, Sweetwater, Florida
  - Fougera Investigational Site, Tampa, Florida
  - Fougera Investigational Site, West Palm Beach, Florida
  - Fougera Investigational Site, Macon, Georgia
  - Fougera Investigational Site, Arlington Heights, Illinois
  - Fougera Investigational Site, New Albany, Indiana
  - Fougera Investigational Site, Plainfield, Indiana
  - Fougera Investigational Site, Louisville, Kentucky
  - Fougera Investigational Site, Lake Charles, Louisiana
  - Fougera Investigational Site, Saint Joseph, Missouri
  - Fougera Investigational Site, Henderson, Nevada
  - Fougera Investigational Site, High Point, North Carolina
  - Fougera Investigational Site, Salem, Oregon
  - Fougera Investigational Site, Hazleton, Pennsylvania
  - Fougera Investigational Site, Upper Saint Clair, Pennsylvania
  - Fougera Investigational Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At Visit 1, eligible subjects were randomized to the Test, Reference or Placebo product in a 1:1:1 ratio using an interactive response technology (IRT) system.
Pre-assignment Details: 927 subjects were screened for study participation, 855 subjects were randomized and included in the statistical analyses.
  29 investigative sites (one with two locations) randomized subjects into the study.
Period: Overall Study
Arm/Group | Test | Reference | Placebo
Started (Randomized (Safety Population)) | 284 | 286 | 285
Modified Intent-to Treat (mITT) (met all inclusion/exclusion criteria, received study treatment, and had a post-Baseline evaluation) | 263 | 266 | 275
Per-Protocol Population (PP) (all randomized subjects who complied with the protocol) | 208 | 209 | 201
Completed | 236 | 235 | 232
Not Completed | 48 | 51 | 53
Not completed — Other | 4 | 3 | 9
Not completed — Withdrawal by Subject | 24 | 18 | 22
Not completed — Significant Worsening of Condition | 0 | 1 | 0
Not completed — Protocol Violation | 2 | 2 | 1
Not completed — Non-Compliance With Study Drug | 0 | 1 | 4
Not completed — Lost to Follow-up | 11 | 13 | 8
Not completed — Lack of Efficacy | 3 | 4 | 5
Not completed — Adverse Event | 4 | 9 | 3
Not completed — Administrative Reasons | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test | Reference | Placebo | Total
Number analyzed (Participants) | 284 | 286 | 285 | 855
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Started (Safety Population)
  Years | 53.5 (14.4) | 53.7 (14.2) | 52.7 (14.2) | 53.3 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Started (Safety Population)
  Participants
    Female | 142 | 129 | 155 | 426
    Male | 142 | 157 | 130 | 429
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Started (Safety Population)
  Participants
    Hispanic or Latino | 172 | 168 | 174 | 514
    Not Hispanic or Latino | 112 | 118 | 111 | 341

OUTCOME MEASURES:

1. Primary Outcome: Treatment Success Assessed by IGA
Description: Proportion of subjects with treatment success (defined as none, minimal or mild disease, a score of 0, 1 or 2 within the treatment area) on the "Investigator's Global Assessment of Disease Severity" (IGA) at the Week 12 visit (Day 85 ± 4 days, End of Study).
Time Frame: Week 12
Population: mITT for superiority versus placebo, PP for equivalence versus Reference
Measure: Number; unit: Percentage of Participants
Arm/Group | Test | Reference | Placebo
Number analyzed (Participants) | 263 | 266 | 275
Percentage of Participants | 60.8 | 63.2 | 56.0
Statistical Analysis 1: Comparison: Test vs Reference; Test type: Equivalence — 90% confidence interval on the difference between the proportions to be within [-20%, +20%]; Yates' corrected confidence interval — p-value not calculated; Risk Difference (RD) = -4.5, 90% CI [-12.6 to 3.6]
Statistical Analysis 2: Comparison: Test vs Placebo; Test type: Superiority — Last Observation Carried Forward (LOCF) for missing efficacy values; p = 0.3520, Cochran-Mantel-Haenszel; stratified by clinical site

2. Secondary Outcome: Disease Severity None or Minimal on IGA
Description: Proportion of subjects with none or minimal disease, a score of 0 or 1 on the IGA at the Week 12 visit (Day 85 ± 4 days, End of Study).
Time Frame: Week 12
Population: mITT
Measure: Number; unit: Percentage of Participants
Arm/Group | Test | Reference | Placebo
Number analyzed (Participants) | 263 | 266 | 275
Percentage of Participants | 17.5 | 22.6 | 16.4
Statistical Analysis 1: Comparison: Test vs Placebo; Test type: Superiority; p = 0.8105, Cochran-Mantel-Haenszel; stratified by clinical site
Statistical Analysis 2: Comparison: Reference vs Placebo; Test type: Superiority; p = 0.0613, Cochran-Mantel-Haenszel; stratified by clinical site

3. Secondary Outcome: Target Site Plaque Elevation, Scaling and Erythema Scores of Less Than or Equal to 1 on the PASI
Description: Proportion of subjects with target site plaque elevation, scaling and erythema scores of less than or equal to 1 (Clear or Almost Clear) on the Psoriasis Area Severity Index (PASI) at the Week 12 visit (Day 85 ± 4 days, End of Study).
Time Frame: Week 12
Population: mITT
Measure: Number; unit: Percentage of Participants
Arm/Group | Test | Reference | Placebo
Number analyzed (Participants) | 263 | 266 | 275
Percentage of Participants | 16.3 | 22.2 | 16.0
Statistical Analysis 1: Comparison: Test vs Placebo; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; stratified by clinical site
Statistical Analysis 2: Comparison: Reference vs Placebo; Test type: Superiority; p = 0.0712, Cochran-Mantel-Haenszel; stratified by clinical site

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit up to approximately 85 days
Arm/Group | Test | Reference | Placebo
All-Cause Mortality (participants affected / at risk) | 0/284 | 0/286 | 0/285
Serious Adverse Events (participants affected / at risk) | 0/284 | 0/286 | 3/285
Other Adverse Events (participants affected / at risk) | 31/284 | 24/286 | 21/285
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test (N=284) | Reference (N=286) | Placebo (N=285)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ischaemic nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Test (N=284) | Reference (N=286) | Placebo (N=285)
Application site dryness (General disorders) | 2 | 4 | 2
Application site erosion (General disorders) | 5 | 4 | 6
Application site erythema (General disorders) | 5 | 5 | 4
Application site pain (General disorders) | 9 | 9 | 10
Application site pruritus (General disorders) | 8 | 4 | 4
Application site rash (General disorders) | 2 | 5 | 1
Nasopharyngitis (Infections and infestations) | 5 | 2 | 3
Sinusitis (Infections and infestations) | 0 | 1 | 3
Headache (Nervous system disorders) | 6 | 2 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Fougera' agreements with its investigators may vary. However, Fougera does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-12-22): https://cdn.clinicaltrials.gov/large-docs/02/NCT02886702/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-26): https://cdn.clinicaltrials.gov/large-docs/02/NCT02886702/SAP_001.pdf